CLINICAL TRIAL: NCT01675115
Title: A Double-Blind, Randomized, Placebo-Controlled, Multi-Center Study to Compare the Functional Outcome and Safety of Treatment With BNG-1 in Combination With Aspirin With That of Aspirin Alone in Ischemic Stroke Recovery
Brief Title: Efficacy of BNG-1 to Treat Acute Ischemic Stroke
Acronym: BNG-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tsong-Hai Lee, Chief of Stroke Center, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNG-1-PIIIB
Record Dates: First submitted 2012-04-02; First posted 2012-08-29 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Traditional Chinese Medication; Aspirin
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BNG-1 plus Aspirin (Active Comparator): BNG-1 3 grams TID plus Aspirin 100mg QD for 4 weeks
  Interventions: Drug: BNG-1
- Aspirin (Sham Comparator): Aspirin 100mg QD for 4 weeks
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: BNG-1 — BNG-1 3 grams TID for 4 weeks
  Arms: BNG-1 plus Aspirin
Drug: Aspirin — Aspirin 100 mg QD for 4 weeks
  Arms: Aspirin

SUMMARY:
The objective of this study is to investigate the efficacy and safety of BNG-1 in patients with ischemic stroke. The efficacy assessment will be based on the functional outcome while the safety will be reviewed by the adverse events and laboratory examinations.

DETAILED DESCRIPTION:
The primary endpoint will be performed on the 12 weeks after study drug administered and will compare the favorable rate between treatment with Aspirin alone and combination treatment with BNG-1 and Aspirin in patients with ischemic stroke. The favorable to therapy will be determined if all of the following occurs: alive, Modified Rankin Scale (MRS) < 3, Barthel Index (BI) >= 60.

Secondary objectives are to compare the following:

1. Compare the favorable rate at one week after study drug administered and the end of treatment (Week 4) and 4 weeks of follow-up (Week 8) of either Aspirin alone or combination treatment with BNG-1 and Aspirin.
2. Compare the mean change in Barthel Index (BI), at each evaluation time-point of either Aspirin alone or combination treatment with BNG-1 and Aspirin.
3. Compare the mean change in National Institute of Health Stroke Scale (NIHSS) at each evaluation time-point of either Aspirin alone or combination treatment with BNG-1 and Aspirin.
4. Compare the Modified Rankin Scale (MRS) at each evaluation time-point of either Aspirin alone or combination treatment with BNG-1 and Aspirin.
5. Compare the change in Extended Glasgow Outcome Scale (GOS-E) at each evaluation time-point of either Aspirin alone or combination treatment with BNG-1 and Aspirin.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders and ages 20 through 65 (subjects are at least 20 years old but not yet 66).
2. Clinical diagnosis of ischemic stroke, causing a measurable neurological deficit.
3. Onset of symptoms of ischemic stroke within 10 days of initiation of treatment with the study drug.
4. Patients have a total National Institutes of Health Stroke Scale (NIHSS) between 8 and 22 inclusive by the time of randomization.
5. Patients have a total Barth Index (BI) less than 60 or Modified Rankin Scale (MRS) at least 3 by the time of randomization.
6. No previous history of stroke or previous stroke with Modified Rankin Scale < 1.
7. Patient must have a CT or MRI examination compatible with the clinical diagnosis of acute ischemic stroke.
8. Signed informed consent from patient or legally authorized representative.

Exclusion Criteria:

1. Patient has only major symptoms that are rapidly improving by the time of randomization.
2. History of stroke within the previous 3 months, exclude TIA.
3. Patient has a CT or MRI scan with evidence of a non-ischemic mechanism, subarachnoid hemorrhage, primary intracerebral or intraventricular hemorrhage.
4. Patients with known or suspected prior intracranial haemorrhage or history of brain injury or brain tumor.
5. Patient had documented history of any atrial fibrillation occurring 6 months before randomization.
6. Hypertension, defined as systolic blood pressure > 185 mmHg or diastolic blood pressure >110 mmHg or requiring aggressive (eg, intravenous antihypertensive) treatment to reduce blood pressure to within these limits.
7. Recurrent peptic ulcer or gastrointestinal bleeding documented by radiographic or endoscopic means within the past 3 months.
8. Pregnant or lactating women or women of childbearing potential who are not practicing reliable birth control.
9. Platelet count less than 100,000 cells/ml.
10. Activated partial thromboplastin time (aPTT) prolongation greater than 2 seconds above the upper limit of normal for local laboratory.
11. International normalized ratio (INR) greater than or equal to 1.4.
12. Uncontrolled hyperglycemia (Sugar AC > 200 mg/dl).
13. History of alcohol or drug abuse in the previous 3 months.
14. History of hypersensitivity or intolerance of study drug or aspirin.
15. Neurological (other than the presenting stroke) or psychiatric conditions that may affect the patient's functional status and/or that may interfere with the patient's assessment.
16. Previously in the BRAIN-Study or participation in a research protocol for investigation of a pharmaceutical agent or innovative invasive procedure within the past 30 days.
17. Any other known clinically significant medical disorder (e.g., a severe comorbid disease or dementia, transient cerebral ischemia, lower gastrointestinal bleeding, bleeding diathesis, hepatorenal diseases, cancer, and AIDS).
18. Patients who have received anticoagulant agents, antiplatelet agents (except Aspirin), thrombolytics with 48-hour before randomization.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Favorable rate | 12 weeks
  Favorite rate: A composite of mortality (alive), modified Rankin Scale < 3, AND Barthel Index (BI)>=60

SECONDARY OUTCOMES:
Favorable rate | 12 weeks
Barthel index | 12 weeks
Modified Rankin Scale | 12 weeks
National Institute of Health Stroke Scale | 12 weeks
Extended Glasgow Outcome Scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tsong-Hai Lee, MD, PhD, Principal Investigator — Chief of Stroke Center, Linkou Chang Gung Memorial Hospital
Locations (1):
- Stroke center, Department of Neurology, Linkou Chang Gung Memorial Hospital, Kweishan, Taoyuan, Taiwan

REFERENCES:
- [Derived] Hsieh CY, Lin HJ. Letter by Hsieh and Lin Regarding Article, "Acute Reperfusion Therapy and Stroke Care in Asia After Successful Endovascular Trials". Stroke. 2015 Aug;46(8):e198. doi: 10.1161/STROKEAHA.115.010253. Epub 2015 Jul 2. No abstract available. PMID 26138124